CLINICAL TRIAL: NCT03836495
Title: The Effect of Bread Fortification With Phosphorus and Lysine on Postprandial Glycaemia and Thermogenesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Omar Obeid, professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BIO-2017-0278
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2019-02

CONDITIONS: Postprandial Hyperglycemia; Energy Expenditure
MeSH Terms: conditions — Hyperglycemia | interventions — Lysine; Phosphorus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- White bread unfortified (WB) (Experimental): bread with no lysine no phosphorus
  Interventions: Dietary Supplement: lysine and phosphorus
- White bread fortified with lysine (WB-L) (Experimental): Bread with lysine
  Interventions: Dietary Supplement: lysine and phosphorus
- White bread fortified with phosphorus (WB-P) (Experimental): bread with phosphorus
  Interventions: Dietary Supplement: lysine and phosphorus
- White bread fortified with lysine and phosphorus (WB-LP) (Experimental): Bread with phosphorus and lysine
  Interventions: Dietary Supplement: lysine and phosphorus

INTERVENTIONS:
Dietary Supplement: lysine and phosphorus — addition of lysine and essential amino acid and/or phosphorus an essential mineral

SUMMARY:
Wheat and wheat derived products are highly consumed around the world. They constitute the major dietary source of protein and energy for many individuals. Wheat contains moderate quantity of low quality protein lacking in some essential amino acids, primarily lysine, thus wheat based diets can't sustain optimal growth, and accordingly should be supplemented with lysine or complemented by another protein source of better quality to match human needs. However, human studies showed that wheat flour fortification with lysine was able to slightly improve growth, namely by increasing weight gain, but it did not however completely reverse growth impairment provoked by the consumption of wheat-based diets.

The investigators developed interest in the role of phosphorus in health and diseased and believe that the modest impact of lysine fortification may due to low phosphorus availability of wheat products. Phosphorus content of cereals is mainly in the form of phytate that is not bioavailable. Supplementing a wheat gluten based diet with a combination of lysine and phosphorus was able to highly amplify the increase in weight gain and energy efficiency of rats as compared to lysine or phosphorus supplementation alone. Phosphorus is an essential mineral known to be directly involved in the production of ATP, which is essential for many metabolic processes including protein synthesis.

The investigators believe that a better approach to enhance the quality of a wheat-based diet is through the supplementation with a combination of both lysine and phosphorus.

The present study is designed to investigate the effect of white flour fortification with lysine and/or phosphorus on sensory properties, postprandial glycaemia and insulinemia, as well as postprandial thermogenesis.

Most specifically, we aim to:

1. Determine the acceptability and assess sensory differences of the fortified breads.
2. Determine the glycemic response after ingestion of the different fortified breads.
3. Evaluate the variation in energy expenditure after the consumption of the fortified breads.

DETAILED DESCRIPTION:
Specific Aim 1: Determine the acceptability and assess sensory differences of the fortified breads.

White wheat flour will be fortified with either lysine, phosphorus, or both lysine and phosphorus. The acceptability of these fortified breads will be tested.

L- Lysine monohydrochloride will be used as the sources of lysine. Potassium phosphate will be used as the source of phosphorus. From previous experience, the addition of potassium phosphate to glucose solution was found to minimally affect the organoleptic properties. Unlike that of sodium phosphate that was not well tolerated by subjects due to development of unfavorable flavor (fishy flavor).

Locally produced white wheat flour (80% extraction) will be purchased and stored at the department. White flour samples will be analyzed for their content of phosphorus according to standard procedures.

Fortification:

Fortification with lysine: 625mg of L-lysine monohydrochloride will be added to 100g of wheat flour, giving a fortification rate of 500mg of lysine (0.5%) in 100g of wheat flour.

Fortification with phosphorus: Phosphorus will be added to white wheat flour in the proportion of 500mg of phosphorus in 100g of white wheat flour, and this will add up to a total of 608mg of phosphorus in 100g of fortified white wheat flour (with 108mg of phosphorus initially present in 100g of unfortified white wheat flour).

Making of breads:

Four different types of bread will be made:

White bread unfortified (WB) White bread fortified with lysine (WB-L) White bread fortified with phosphorus (WB-P) White bread fortified with lysine and phosphorus (WB-LP)

Acceptability of the four different breads:

Bread samples will be tested for acceptability. Panelists (n= 60) will be recruited based on their willingness to participate in the study and their consumption of Arabic bread.

Panelists will be asked to fill a questionnaire and to rate the served samples on a 9-point hedonic scale with 1 representing dislike extremely and 9 representing like extremely for overall acceptability, acceptability of appearance, texture and taste. The order of presentation of the samples will be counterbalanced.

Sensory evaluation of the four different breads:

Panelists (n=24) who are regular consumers of white bread will be recruited to assess any sensory differences between experimental samples of the white bread control and the three white breads supplemented with lysine and/or phosphorus. The triangle test will be used in the difference tests.

All subjects will be asked to sign human subjects consent forms and answer demographic information. Demographic information that will be requested will be: 1) age, 2) gender, 3) frequency of bread consumption, 4) type of bread typically consumed, and 5) what factors influence the panelists' bread purchase.

Twenty four panelists will participate in three triangle test, comparing the white bread control vs. each of the three experimental samples in each test. In the session, subjects will be debriefed about a) the products they will consume, b) the procedures for the testing, c) instructions on how to sample the beverages, and d) how to use the score card. All samples will be presented in a random, balanced order.

Mineral and carbohydrate content of bread:

Phosphorus content of the breads will be determined.

Specific Aim 2: Determine the glycemic response following the consumption of the different fortified breads.

In this experiment, healthy subjects (n=12) will be recruited and asked to maintain their regular dietary and physical activity habits during the entire study course, avoid alcohol consumption as well as any unusual strenuous exercise 24 hours prior to the study.

Exclusion criteria: any significant medical diseases; pregnancy or lactation; regular use of medication that affects body weight; a weight loss of 3% or more in the preceding 3 months.

Following a 12 hour (overnight) fast, subjects will be taken to the testing facility [Faculty of Agriculture and Food Sciences/Department of Nutrition or the Central research unit (CRU)/ American University Hospital] where anthropometric measurements (height, weight) will be taken. A catheter will be inserted for blood withdrawal.

Postprandial glycemic response after consumption of the four fortified breads will be determined.

A crossover design will be used in which each subject will undertake 4 visits in a random order over 4 different days, the difference between the visits being the type of bread to be consumed.

In brief, overnight fasted subjects will be given the bread (50 g of carbohydrate) to ingest within 10-15 min and drink 250 ml of water. Blood samples will be taken immediately before the meal and at 15, 30, 45, 60, 90 and 120 minutes after meal ingestion. Blood will be withdrawn by a trained practitioner and will be used for the determination of glucose.

Glucose area under the curve (AUC) will be calculated. In addition, mineral and several metabolites content of the blood will be measured (glucose, total phosphorus, triglycerides, insulin and GLP-1).

Specific Aim 3: Evaluate the variation in Energy Expenditure after the consumption of the fortified breads.

Subject recruitment: 16 healthy subjects in total will be recruited. 14 subjects will be required in order to be able to detect significance at the level of 0.05, using a 25% difference between treatments and 90% power. But, a total number of 16 subjects will be recruited in order to allow for the loss which might take place due to the dropping out.

Inclusion criteria: 16 subjects (BMI between 20 and 25) will be recruited. Efforts will be made to age and gender match subjects (balanced number of males and females in each group). Subjects are appropriate if they are in the age range between 18 and 60. Women who are in the reproductive age will be studied at the first half of their menstrual cycle, because estrogen is known to affect the energy expenditure. Postmenopausal women taking hormonal replacement therapy will be excluded. Subjects should have: Cr <1mg/dl for women and <1.2mg/dl for men and GFR >60 ml/min/1.73m2.

ELIGIBILITY:
Inclusion Criteria:

* Efforts will be made to age and gender match subjects (balanced number of males and females in each group). Subjects are appropriate if they are in the age range between 18 and 60. Women who are in the reproductive age will be studied at the first half of their menstrual cycle, because estrogen is known to affect the energy expenditure. Postmenopausal women taking hormonal replacement therapy will be excluded. Subjects should have: Cr <1mg/dl for women and <1.2mg/dl for men and GFR >60 ml/min/1.73m2.

Exclusion Criteria:

* Subjects with diabetes, cardiovascular, cerebrovascular, pulmonary, hepatic, renal, endocrinological (PTH), or any significant medical disease will be excluded.
* Pregnant and lactating women.
* Subjects on regular use of medication that affects body weight and/or having a weight loss of 3% or more in the preceding 3 months.
* Subjects with: Cr >1mg/dl for women and >1.2mg/dl for men and GFR<60 ml/min/1.73m2.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemia | 120 min
  postprandial blood glucose level
Energy expenditure | 240 min
  Postprandial energy expenditure

CONTACTS AND LOCATIONS:
Overall Officials: Omar Obeid, PhD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided